CLINICAL TRIAL: NCT03893162
Title: Gut Feeling: Understanding the Mechanisms Underlying the Antidepressant Properties of Probiotics
Acronym: PROMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PROMEX
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
Keywords: probiotic; depression; microbiome; bacteria
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-strain probiotic "BioKult" (Experimental): 4 capsules daily for 8 weeks
  Interventions: Dietary Supplement: Multi-strain probiotic
- Placebo (Placebo Comparator): 4 capsules daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-strain probiotic — The intervention in this study is a multi-strain probiotic which contains:
  Bacillus subtilis, Bifidobacterium bifidum, Bifidobacterium breve, Bifidobacterium infantis, Bifidobacterium longum, Lactobacillus acidophilus, Lactobacillus delbrueckii ssp. bulgaricus, Lactobacillus casei, Lactobacillus plantarum, Lactobacillus rhamnosus, Lactobacillus helveticus, Lactobacillus salivarius, Lactococcus lactis ssp. lactis, Streptococcus thermophilus.
  Each capsule contains minimum 2 billion live microorganisms per capsule, equivalent to 10 billion live microorganisms per gram.
  Other Names: "BioKult"
  Arms: Multi-strain probiotic "BioKult"
Other: Placebo — Visually identical capsules in identical packaging containing no active bacteria.
  Arms: Placebo

SUMMARY:
Previous research has suggested that probiotics can improve depressive symptoms in patients with Major Depressive Disorder (MDD), particularly when used in addition to antidepressants. The aim of this exploratory pilot study is to improve the investigator's understanding of the mechanisms underlying these effects. This study will assess the effects of an 8-week double-blind placebo-controlled probiotic intervention on the gut microbiome, inflammatory marker levels, brain activity and neurotransmitter levels in patients with MDD and their relationship to changes in mood. This study will also recruit a group of demographically-matched healthy controls for gut microbiome comparison with the MDD group (non-interventional).

ELIGIBILITY:
Inclusion criteria for MDD participants:

* aged 18-55;
* currently in a depressive episode according to DSM-5 criteria, who are currently on antidepressant treatment but remain symptomatic (HAM-D17 score >13);
* on stable treatment regimen of an approved treatment for at least 6 weeks;
* non-smokers;
* for participants willing to take part in the neuroimaging component: right-handed, no contraindications, non-claustrophobic, weight <126kg;

Exclusion criteria for MDD participants:

* eating disorder, bipolar disorder, schizophrenia or psychotic symptoms;
* substance dependence in the past year, except for caffeine;
* active suicidal ideation;
* use of probiotic supplements in the past 2 weeks, or regular use of a probiotic;
* use of antibiotics in the past 12 weeks;
* history of allergic reaction to any of the components of BioKult;
* history of history of a systemic medical illness;
* current presence of significant GI problems or disease or history of major GI surgery;
* pregnancy or breastfeeding;
* following a dietary regimen unrepresentative of the general population (e.g. fasting or following a specific diet);
* regular/current use of antacids, proton pump inhibitors, laxatives, antidiarrheals;

Inclusion criteria for Healthy Volunteers:

* Aged 18-55;
* No current or historic presence of depression, other psychiatric disorder or substance dependence
* No history of a systemic medical illness;
* No family history of psychiatric disorder;
* Non-smoker;
* Not used probiotic supplements in the past 2 weeks, nor regular use of a probiotic;
* Not used antibiotics in the past 12 weeks;
* No current presence of gastrointestinal disease, or history of major GI surgery;
* No reported regular/current use of antacids, proton pump inhibitors, laxatives, antidiarrheals;
* pregnancy or breastfeeding;
* not currently following a dietary regimen or dietary restrictions unrepresentative of the general population (e.g. fasting or following a specific diet);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
gut microbiota in MDD | baseline
  species diversity and abundance at the level of organisational taxonomic units (OTUs) will be measured with 16S ribosomal RNA (rRNA) sequencing
differences in gut microbiota between MDD and healthy volunteers | baseline
  species diversity and abundance at the level of OTUs will be measured with 16SrRNA-based sequencing and compared between the two groups
gut microbiota changes in MDD following probiotic intervention and their correlation to change in depressive symptoms | change from baseline to week 8
  species diversity and abundance at the level of OTUs will be measured with 16SrRNA-based sequencing and depressive symptoms will be measured with the Inventory of Depressive Symptomatology Self-Report (IDS-SR) and the Hamilton Depression Rating Scale (HAM-D17)

SECONDARY OUTCOMES:
Neurotransmitters | change from baseline to week 8
  levels of glutamate and gamma-aminobutyric acid (GABA) will be measured with Magnetic Resonance Imaging (MRS)
Blood | change from baseline to week 8
  levels of tumor necrosis factor (TNF-a), interleukins IL-1β, IL-6, IL-17, and C-reactive protein (CRP) will be measured
Brain activity | change from baseline to week 8
  measured with functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: James M Stone, MBBS PhD FRCPsych, Principal Investigator — Institute of Psychiatry Psychology and Neuroscience, King's College London
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Derived] Nikolova VL, Cleare AJ, Young AH, Stone JM. Exploring the mechanisms of action of probiotics in depression: Results from a randomized controlled pilot trial. J Affect Disord. 2025 May 1;376:241-250. doi: 10.1016/j.jad.2025.01.153. Epub 2025 Feb 7. PMID 39924003
- [Derived] Nikolova VL, Cleare AJ, Young AH, Stone JM. Acceptability, Tolerability, and Estimates of Putative Treatment Effects of Probiotics as Adjunctive Treatment in Patients With Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Aug 1;80(8):842-847. doi: 10.1001/jamapsychiatry.2023.1817. PMID 37314797